CLINICAL TRIAL: NCT04822376
Title: Phase IIa Pilot Study Evaluating the Efficacy of a Monoclonal Antibody and Vaccine-based Post-exposure Prophylaxis Strategy in High-risk Contact Cases of Ebola Virus Disease Infection
Brief Title: Prophylaxis Vaccine Antibodies Ebola
Acronym: PROVAE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 0006S
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — ansuvimab

STUDY DESIGN:
Intervention Model Description: Efficacy trial : Exploratory, non-comparative, unblinded trial with Mab at D0 and vaccine at W6.
  Immunological ancillary study : Exploratory, controlled, comparative, non-randomized, 2-group, unblinded study comparing Mab at D0 and vaccine at W6 for high-risk contacts with vaccine at D0 for vaccinated contacts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High risk arm (Experimental): Mabs at day 0 and vaccine at week 6
  Interventions: Drug: ansuvimab; Biological: Ervebo
- High risk arm (Immunological ancillary study) (Experimental): Mabs at day 0 and vaccine at week 6
  Interventions: Drug: ansuvimab; Biological: Ervebo
- Control arm (Immunological ancillary study) (Active Comparator): Vaccine at day 0 for contacts eligible for vaccination
  Interventions: Biological: Ervebo

INTERVENTIONS:
Drug: ansuvimab — Human monoclonal antibody to Zaire strain GP (EBOV GP)
  Other Names: mab114
  Arms: High risk arm; High risk arm (Immunological ancillary study)
Biological: Ervebo — Ebola Zaire vaccine (rVSV∆G-ZEBOV-GP, live, attenuated) ≥ 72 million PFU, composed of the Indiana strain of recombinant vesicular stomatitis virus (rVSV) with a deletion of the envelope glycoprotein (G) of VSV replaced by the surface glycoprotein (GP) of the Kikwit 1995 strain of Ebola virus Zaire (ZEBOV)
  Other Names: VSV-ZEBOV

SUMMARY:
* Three measures are currently being implemented to control Ebola outbreaks:

  * Monitoring of contacts
  * Isolation and treatment of sick people
  * Vaccination of the population in high-risk areas.
* In contacts with high viral exposure and therefore a high risk of incubation and rapid expression of infection, the r-VSV-ZEBOV vaccine does not provide adequate protection because vaccine antibody production is effective 6 to 10 days after administration.
* Specific monoclonal antibodies (Mab) from the Regeneron and mAb114 research specialties have been shown to be effective in reducing mortality in patients with Ebola virus disease (EVD).
* Their use in a single parenteral administration and good tolerability make them candidates for use in post-exposure prophylaxis (PEP) in individuals at high risk of viral exposure.
* A comprehensive strategy for the protection of high-risk contacts must therefore be implemented, including the vaccine and the Mabs, to ensure both immediate and prolonged protection. Indeed, the efficacy of the vaccine is likely to be diminished when co-administered with Mabs, as both strategies share the same viral target (the GP envelope glycoprotein) and the vaccine is replicative (and therefore may be inhibited by Mabs).

PROVAE aim to evaluate the effectiveness of a comprehensive strategy to prevent transmission of MVE in contacts at high risk of infection, including (i) post-exposure prophylaxis with Mabs and (ii) vaccination with r-VSV-ZEBOV.

ELIGIBILITY:
The inclusion criteria for the efficacy trial are:

* Have had, within the previous 72 hours, a high-risk contact with an Ebola patient confirmed by RT-PCR;
* Be 18 years of age or older at the time of inclusion;
* Have no symptoms of EVD;
* Give consent to participate in the efficacy trial;
* Agree not to participate in any other therapeutic or vaccine study until the end of the trial follow-up.

The criteria for non-inclusion in the efficacy trial are:

* Have a history of EVD (self-report);
* Have been vaccinated with ERVEBO prior to the start of the study;
* Have participated in another therapeutic or vaccine study within 15 days prior to inclusion.

Inclusion criteria for the immunology ancillary study are:

High Risk Arm:

* Be included in the efficacy trial;
* Be available for extended follow-up as specified in the protocol;
* Specifically consent to the immunology ancillary study.

Control arm:

* Be 18 years of age or older at the time of inclusion;
* Have no symptoms of EVD;
* Eligible for ERVEBO vaccination according to national program criteria;
* Be available for extended follow-up as specified in the protocol;
* Consent specifically for the ancillary immunology study.

The criteria for non-inclusion in the immunologic ancillary study are:

* All efficacy trial non-inclusion criteria;
* HIV positive;
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-10-17 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy | Week 3
  Proportion of participants with negative RT-PCR
Immunological ancillary study | 6 months after vaccination
  Anti-GP IgG level (FANG reference technique)

SECONDARY OUTCOMES:
Tolerance | Day 7 post-PEP and day 7 post-vaccination
  Estimating adverse effects
Lost of follow-up | Week 6
  Lost of follow-up rate
Humoral immune response | 1 and 3 months after vaccination
  Anti-GP IgG level (FANG reference technique)
Neutralizing antibodies | 1, 3 and 6 months after vaccination
  Neutralizing antibodies level

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Traitement Ebola de N'Zerekore, N'Zerekore, Guinea